CLINICAL TRIAL: NCT05166239
Title: Hepatic Arterial Infusion Chemotherapy Combine With Lenvatinib and PD-1 Inhibitors for Advanced Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis.
Brief Title: HAIC Combine With Lenvatinib and PD-1 Inhibitors for Advanced HCC With PVTT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Wang, MD, Professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAIC-Cola
Record Dates: First submitted 2021-11-26; First posted 2021-12-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Thrombosis
Keywords: Hepatocellular Carcinoma; Portal Vein Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC-Cola group (Experimental): Hepatic arterial chemotherapy consisted of infusions of oxaliplatin (35 mg/m2 for 2 hours), followed by 5-fluorouracil (600 mg/m2 for 22 hours) on day1-3 every 4 weeks. 12/8 mg (weight ≥ 60kg / < 60 kg) of Lenvatinib once daily after HAIC. PD-1 inhibitors injection intravenously or percutaneously before 24h of HAIC every 4 week.
  Interventions: Procedure: HAIC; Drug: Lenvatinib 1; Drug: PD-1 Inhibitors
- Cola group (Active Comparator): 12/8 mg (weight ≥ 60kg / < 60 kg) of Lenvatinib once daily. PD-1 inhibitors injection intravenously or percutaneously every 4 week.
  Interventions: Drug: Lenvatinib 2; Drug: PD-1 inhibitors 2

INTERVENTIONS:
Procedure: HAIC — Hepatic arterial chemotherapy consisted of infusions of oxaliplatin (35 mg/m2 for 2 hours), followed by 5-fluorouracil (600 mg/m2 for 22 hours) on day1-3 every 4 weeks.
  Arms: HAIC-Cola group
Drug: Lenvatinib 1 — 12/8 mg (weight ≥ 60kg / < 60 kg) of Lenvatinib once daily after HAIC.
  Arms: HAIC-Cola group
Drug: PD-1 Inhibitors — PD-1 inhibitors injection intravenously or percutaneously before 24h of HAIC every 4 week.
  Other Names: PD-1
  Arms: HAIC-Cola group
Drug: Lenvatinib 2 — 12/8 mg (weight ≥ 60kg / < 60 kg) of Lenvatinib once daily.
  Arms: Cola group
Drug: PD-1 inhibitors 2 — PD-1 inhibitors injection intravenously or percutaneously every 4 week.
  Arms: Cola group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of hepatic arterial infusion chemotherapy combined with Lenvatinib and PD-1 inhibitors compared to Lenvatinib plus PD-1 inhibitors for advanced hepatocellular carcinoma (HCC) with portal vein tumor thrombosis (PVTT).

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC) can significantly improve the local drug concentration in liver compared to systemic chemotherapy. The efficacy of HAIC for hepatocellular (HCC), cholangiocarcinoma, gallbladder, and colorectal carcinoma liver metastasis has been proved by many published studies. HAIC with oxaliplatin and 5-fluorouracil could significantly prolong survival time for HCC patients with portal vein tumor thrombosis (PVTT). Lenvatinib, as a new oral anti-neovascularity inhibitor, was proved to have similar efficacy in HCC patients compared to sorafenib in REFLECT study. The sub-group analysis showed that the median overall survival (OS) in Lenvatinib group was significantly longer that sorafenib group in Chinese HCC patients. Recently, the programmed death-1 (PD-1) inhibitors alone or combined with targeted therapy was explored and confirmed to be effective for advanced HCC, with the median progression-free survival (PFS) and median OS of 2.1-5.6 months and 14.4-22.1 months, resepectively. Thus, the investigators carried out this prospective controlled trial to compare the efficacy and safety of HAIC combined with Lenvatinib and PD-1 inhibitors and Lenvatinib and PD-1 inhibitors for advanced HCC with PVTT.

Total 66 subjects will be recruited in this trial, each group of 33 subjects in treatment group (HAIC-Cola group) and control group (Cola group). The primary endpoint is six-month progression-free survival rate, and the secondary endpoints are OS, overall response rate (ORR), PFS, time-to-progression (TTP) and safety. The safety evaluation will be carried out according to the standard of adverse reaction classification (Common Terminology Criteria for Adverse Events, CTCAE v5.0).

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: >18 years old and≤75 years old, both men and women.
2. All subjects must have advanced hepatocellular carcinoma with portal vein tumor thrombosis confirmed by pathological or clinical diagnosis.
3. One measurable lesion at least.
4. ECOG PS 0-1 before 1 week of treatment begnining.
5. Child-Pugh class A; ALBI class 1-2.
6. Systemic-cheomtherapy-naive and HAIC-naive.
7. BCLC C stage with PVTT (Vp1 - Vp4).
8. Without distant metastasis.
9. Patients who are expected to live more than 3 months.
10. Subjects must volunteer to participate in the study, signed informed consent, and were able to comply with the program requirements of visits and related procedures.
11. Patients with laboratory values that meet the following criteria:

    1. Hemoglobin≥90 g/L;
    2. Neutrophile granulocytes≥1.5×109/L;
    3. Platelet count≥75×109/L;
    4. Albumin≥30 g/L;
    5. Total serum bilirubin ≤ 2 times upper limits of normal;
    6. AST and ALT ≤ 5 times upper limits of normal;
    7. Serum creatinine ≤ 1.5 times upper limits of normal;
    8. Alkaline phosphatase ≤ 5 times upper limits of normal;
    9. Prothrombin time or international normalized ratio ≤ 1.5 times upper limits of normal, activated partial thromboplastin time (APTT) ≤ 1.5×ULN.

Exclusion Criteria:

1. Fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma confirmed by histology or cytology.
2. History of malignant tumor, excluding the following cases:
3. Allergic to contrast agent.
4. Allergic to oxaliplatin.
5. History of usage of immune inhibitor drug within 14 days before the injection of PD-1 inhibitors, except nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (no more than 10 mg/day of prednisolone or other corticosteroids with equivalent physiological doses).
6. Factors influenced oral Lenvatinib, such as inability to swallow, chronic diarrhea and intestinal obstruction, or other conditions that significantly affect the administration and absorption of the drug.
7. Allergic to Lenvatinib, PD-1 inhibitors, and other mono-colonal antibodies.
8. Vaccination with live attenuated vaccine within 4 weeks before the first dose or planned during the study period.
9. Peripheral neuropathy> Grade 1.
10. History of active autoimmune disease or autoimmune disease.
11. History of other malignant tumor, except for radically treated basal cell, squamous cell skin cancer, or cervical carcinoma in situ.
12. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) .
13. Clinically significant cardiovascular disease, including, but not limited to, acute myocardial infarction, severe/unstable angina or prior coronary artery bypass surgery, congestive heart failure (NYHA >2), poorly controlled arrhythmias or arrhythmias requiring pacemaker therapy, hypertension not controlled by medication (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) within the past 6 months.
14. Abnormal coagulation function (INR>1.5 or APTT>1.5×ULN) , have bleeding tendency, or are receiving thrombolytic therapy, anticoagulation therapy or antiplatelet therapy, etc..
15. History of inherited or acquired bleeding and thrombotic tendency, such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc..
16. History of significant coughing up blood 2 months before entering the study, or the daily volume of hemoptysis reached 2.5 ml or more.
17. Patients at risk of gastrointestinal bleeding, including the following:

    1. There are active peptic ulcer lesions.
    2. Those who have a history of melena and hematemesis within 3 months.
    3. For fecal occult blood (+) or (+/-), it is necessary to recheck the stool routine within 1 week. Those who still (+) or (+/-) must undergo gastroscopy. If there is ulcer, bleeding disease, and the treating physician believes that there is a potential risk of bleeding.
18. History of thrombosis and/or embolism within 6 months of the start of treatment.
19. Complicated infections requiring drug intervention (such as intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks before the first treatment, or unexplained fever >38.5°C during the screening period/before the first administration.
20. Participated in any other clinical research within 4 weeks before the first treatment.
21. History of psychotropic drug abuse or drug use.
22. Other serious physical, mental illnesses or laboratory abnormalities, which may increase the risk of participating in the research or interfere with the results of the research, and those who the researcher believes are not suitable for participating in this research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
6-month progression-free survival rate | From the date of treatment begining to the date of 6 months after the treatment begining.
  Proportion of patients with 6- month progression-free survival after treatment begining in all patients.

SECONDARY OUTCOMES:
Overall survival | From date of treatment beginning until the date of death from any cause, assessed up to 100 months.
  The time from treatment initiation to death due to any cause
Objective survival rate | Evaluation of tumor burden based on mRECIST criteria through study completion, an average of once per 3 months.
  The proportion of participants in the analysis population who have complete response (CR) or partial response (PR) determined by investigators using mRECIST criteria at any time during the study.
Progression-free survival | From date of treatment beginning until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  The time from treatment initiation to the first documented disease progression or death due to any cause, whichever occurs firstly.
Time to progression | Evaluation of tumor burden based on mRECIST criteria until first documented progress, assessed up to 100 months.
  Time to progression is defined as time from treatment initiation to radiological progression.
Number of patients with treatment-related adverse events | Through study completion, an average of once per 1 month.
  Number of patients with AE, treatment-related AE (TRAE), serious adverse event (SAE) assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Wang, MD, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking Univerisity Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Background] Llovet JM, Montal R, Villanueva A. Randomized trials and endpoints in advanced HCC: Role of PFS as a surrogate of survival. J Hepatol. 2019 Jun;70(6):1262-1277. doi: 10.1016/j.jhep.2019.01.028. Epub 2019 Mar 31. PMID 30943423
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Boussiotis VA. Molecular and Biochemical Aspects of the PD-1 Checkpoint Pathway. N Engl J Med. 2016 Nov 3;375(18):1767-1778. doi: 10.1056/NEJMra1514296. No abstract available. PMID 27806234
- [Background] Ma W, Gilligan BM, Yuan J, Li T. Current status and perspectives in translational biomarker research for PD-1/PD-L1 immune checkpoint blockade therapy. J Hematol Oncol. 2016 May 27;9(1):47. doi: 10.1186/s13045-016-0277-y. PMID 27234522
- [Background] Jia Y, Zeng Z, Li Y, Li Z, Jin L, Zhang Z, Wang L, Wang FS. Impaired function of CD4+ T follicular helper (Tfh) cells associated with hepatocellular carcinoma progression. PLoS One. 2015 Feb 17;10(2):e0117458. doi: 10.1371/journal.pone.0117458. eCollection 2015. PMID 25689070
- [Background] Finn RS, Ryoo BY, Merle P, Kudo M, Bouattour M, Lim HY, Breder V, Edeline J, Chao Y, Ogasawara S, Yau T, Garrido M, Chan SL, Knox J, Daniele B, Ebbinghaus SW, Chen E, Siegel AB, Zhu AX, Cheng AL; KEYNOTE-240 investigators. Pembrolizumab As Second-Line Therapy in Patients With Advanced Hepatocellular Carcinoma in KEYNOTE-240: A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2020 Jan 20;38(3):193-202. doi: 10.1200/JCO.19.01307. Epub 2019 Dec 2. PMID 31790344
- [Background] Gunda V, Gigliotti B, Ashry T, Ndishabandi D, McCarthy M, Zhou Z, Amin S, Lee KE, Stork T, Wirth L, Freeman GJ, Alessandrini A, Parangi S. Anti-PD-1/PD-L1 therapy augments lenvatinib's efficacy by favorably altering the immune microenvironment of murine anaplastic thyroid cancer. Int J Cancer. 2019 May 1;144(9):2266-2278. doi: 10.1002/ijc.32041. Epub 2019 Jan 24. PMID 30515783
- [Background] Kato Y, Tabata K, Kimura T, Yachie-Kinoshita A, Ozawa Y, Yamada K, Ito J, Tachino S, Hori Y, Matsuki M, Matsuoka Y, Ghosh S, Kitano H, Nomoto K, Matsui J, Funahashi Y. Lenvatinib plus anti-PD-1 antibody combination treatment activates CD8+ T cells through reduction of tumor-associated macrophage and activation of the interferon pathway. PLoS One. 2019 Feb 27;14(2):e0212513. doi: 10.1371/journal.pone.0212513. eCollection 2019. PMID 30811474
- [Background] Makker V, Rasco D, Vogelzang NJ, Brose MS, Cohn AL, Mier J, Di Simone C, Hyman DM, Stepan DE, Dutcus CE, Schmidt EV, Guo M, Sachdev P, Shumaker R, Aghajanian C, Taylor M. Lenvatinib plus pembrolizumab in patients with advanced endometrial cancer: an interim analysis of a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2019 May;20(5):711-718. doi: 10.1016/S1470-2045(19)30020-8. Epub 2019 Mar 25. PMID 30922731
- [Background] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452
- [Background] Song Y, Wu J, Chen X, Lin T, Cao J, Liu Y, Zhao Y, Jin J, Huang H, Hu J, Luo J, Zhang L, Xue H, Zhang Q, Wang W, Chen C, Feng J, Zhu J. A Single-Arm, Multicenter, Phase II Study of Camrelizumab in Relapsed or Refractory Classical Hodgkin Lymphoma. Clin Cancer Res. 2019 Dec 15;25(24):7363-7369. doi: 10.1158/1078-0432.CCR-19-1680. Epub 2019 Aug 16. PMID 31420358
- [Background] Nie J, Wang C, Liu Y, Yang Q, Mei Q, Dong L, Li X, Liu J, Ku W, Zhang Y, Chen M, An X, Shi L, Brock MV, Bai J, Han W. Addition of Low-Dose Decitabine to Anti-PD-1 Antibody Camrelizumab in Relapsed/Refractory Classical Hodgkin Lymphoma. J Clin Oncol. 2019 Jun 10;37(17):1479-1489. doi: 10.1200/JCO.18.02151. Epub 2019 Apr 30. PMID 31039052
- [Background] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638
- [Background] Zhu H, Yang X, Zhao Y, Yi C. Efficacy of anti-PD-1 antibody SHR-1210 as second-line treatment in hepatocellular carcinoma patient with sorafenib resistance: A case report. Medicine (Baltimore). 2019 May;98(20):e15755. doi: 10.1097/MD.0000000000015755. PMID 31096541
- [Background] Zhang Z, Zhou Y, Hu K, Li Z, Wang Z, Huang Y. Complete response of early stage hepatocellular carcinoma in a patient treated with combination therapy of camrelizumab (SHR-1210) and apatinib. Dig Liver Dis. 2019 Oct;51(10):1488-1490. doi: 10.1016/j.dld.2019.07.005. Epub 2019 Aug 7. No abstract available. PMID 31401020
- [Background] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Hodi FS, Ballinger M, Lyons B, Soria JC, Nishino M, Tabernero J, Powles T, Smith D, Hoos A, McKenna C, Beyer U, Rhee I, Fine G, Winslow N, Chen DS, Wolchok JD. Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST): Refining Guidelines to Assess the Clinical Benefit of Cancer Immunotherapy. J Clin Oncol. 2018 Mar 20;36(9):850-858. doi: 10.1200/JCO.2017.75.1644. Epub 2018 Jan 17. PMID 29341833